CLINICAL TRIAL: NCT03500029
Title: The Study About Mechanism of Transcranial Magnetic Stimulation Treatment of Patients With Depression Using Multimodal Magnetic Resonance Imaging
Brief Title: The Study About Mechanism of Transcranial Magnetic Stimulation Treatment of Depression Using Medical Imaging
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Chenwang Jin, chief physician, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JIN1115
Record Dates: First submitted 2018-02-07; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Depression
Keywords: Depression; Transcranial magnetic stimulation(TMS); Resting-state functional MRI(fMRI)
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation; Antidepressive Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TMS treatment group (Experimental): In the Transcranial magnetic stimulation (TMS) treatment group patients with severe depression receive rTMS treatment without drug treatment.
  Interventions: Radiation: Transcranial magnetic stimulation (TMS)
- medication group (Active Comparator): In the medication group patients with severe depression are treated with anti-depressants.
  Interventions: Drug: antidepressants
- healthy control group (No Intervention): The control group don't accept intervention and treatment.

INTERVENTIONS:
Radiation: Transcranial magnetic stimulation (TMS) — TMS treatment group is treated with TMS for 20-40 minutes a time, 5 times a week. The stimulation parameters were 20 Hz and 80% MT. Each stimulation continues for 2 seconds, and the interval time of stimulation is 58 seconds.
  Arms: TMS treatment group
Drug: antidepressants — Medication group is treated with anti-depression for 6 weeks. The drugs and their doses belong to the first-line treatment for depression in the current guideline .
  Arms: medication group

SUMMARY:
Depression is the most common psychiatric condition and a important public health concern in society. But medications for depression don't work as well as people expected and cause serious side-effects. Transcranial magnetic stimulation (TMS) is a noninvasive electrical stimulation treatment for depression, which has been approved by the FDA and added to the Guidelines for the Treatment of Depression in China. Despite the effect of the treatment is clear ,the TMS target,the neural circuit which plays a role in TMS and its mechanism remain unknown now. TBS target and effective site may be not in the same position. A large number of previous studies demonstrate the advantages and application prospects of different techniques of magnetic resonance (MR)in the study of pathogenesis of depression. Based on the results of previous research supported by the National Natural Science Foundation of China,the National Key Technology Research and Development Program of China during the "10th Five-Year Plan" and New Health Care and New technology. project team puts forward the idea of joint use of brain structure imaging of MR ,Diffusion Tensor Imaging (DTI) and resting-state functional MRI (fMRI) with different analysis methods to conduct a comprehensive study. The study is focused on the effects of TBS treatment on brain structure network, fiber connectivity network and functional connectivity network ,and nodes affected by it. Then we make further investigation about the mechanism of TMS treatment. The research will provide not only help for studying the pathogenesis of depression but also more reliable targets of next TMS treatment.

DETAILED DESCRIPTION:
The advantages of 3D T1 WI are thin slice scan，no interval, scanning fast and three-dimension reconstruction in any orientation compared with 2D SE. It is not easy to miss small lesions, and shows normal anatomy and lesions more objectively and more accurately.

Doppler tissue imaging (DTI) can reflect white matter fiber so that can be used to determine whether the various diseases affect nerve cell connections.

Arterial spin labeling (ASL) is non-drug perfusion imaging and completely noninvasive technology which can reflect brain perfusion better.

Resting-state functional MRI (fMRI) is used to located the abnormal brain regions whose activity is consistent with dorsolateral prefrontal cortex (DLPFC) by the abnormal resting spontaneous brain activity in patients with depression and the abnormal functional connectivity network.

ELIGIBILITY:
Inclusion Criteria:

TMS treatment group and medication group:

1. Hospitalized patients or outpatients which meet Clinical diagnosis of depression such as international Classification of diseases-10( ICD-10) which is the diagnostic criteria of unipolar depression;Scores of Hamilton Depression Scale (HAMD) ≥ 18 points, scores of clinical total impression scale (CGI)≥ 3 points, and without severe suicidal tendency;
2. 18-60 years old, male or female;
3. Physical and laboratory examination, electrocardiogram(ECG),and electroencephalogram (EEG) with no abnormal changes;
4. No serious or unstable cerebrovascular, liver, kidney, endocrine, blood and other somatic diseases;
5. The patient or the legal guardian should sign a written informed consent after fully understanding the research content of this study.

Healthy control group:

1. 18-60 years old, male or female;
2. Physical and laboratory examination, electrocardiogram(ECG),and electroencephalogram (EEG) with no abnormal changes;
3. No serious or unstable heart, liver, kidney, endocrine, blood and other somatic diseases;
4. Subjects or their legal guardians sign written informed consents after fully understanding the research contents of this study.

Exclusion Criteria:

1. Mental disorders caused by organic diseases such as brain tumors;
2. Serious somatic diseases, severe suicidal tendency and pacemakers;
3. Secondary depressive disorder, psychotic depression or bipolar disorder caused by drugs;
4. Antidepressants or psychoactive drugs were taken one month before enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale-17(HAMD-17) | Difference at HAMD-17 between day 1，week 2 and week 4.
  HAMD-17 are to evaluate the severity degree of depression and the clinical effectiveness for treatment of depression.HAMD-17 scores range in 0-52 points.Total score which is between 7 and 16 means that volunteer may be with depression.Total score which is between 17 and 23 means that volunteer certainly is with depression.Total score which is more than 23 means that volunteer is with severe depression.
Multimodal Magnetic Resonance Imaging | Difference at Multimodal Magnetic Resonance Imaging between day 1,week 2 and week 4.
  Multimodal Magnetic Resonance Imaging include 3D-T1, ASL, DTI, resting-state functional MRI, etc.these show the Brain changes.

SECONDARY OUTCOMES:
Clinical Global Impression.(CGI) | Difference at CGI between day 1，week 2 and week 4.
  CGI is to evaluate the severity degree of depression to estimate whether patients are in accordance with inclusion criteria which concludes severty of illness (si),global improvement (gi) and efficacy index (ei).Si scores range in 0-7 points.Gi scores range in 0-7 points.Ei scores range in 0-4.00 points.
Wisconsin Card Sorting Test (WCST) | Difference at WCST between day 1,week 2 and week 4.
  WCST is to to evaluate the cognitive function of volunteers.Total score which is less 69 means that volunteer suffers from mental deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Chenwang Jin, doctorate, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bora E, Fornito A, Pantelis C, Yucel M. Gray matter abnormalities in Major Depressive Disorder: a meta-analysis of voxel based morphometry studies. J Affect Disord. 2012 Apr;138(1-2):9-18. doi: 10.1016/j.jad.2011.03.049. Epub 2011 Apr 20. PMID 21511342
- [Result] Chase HW, Nusslock R, Almeida JR, Forbes EE, LaBarbara EJ, Phillips ML. Dissociable patterns of abnormal frontal cortical activation during anticipation of an uncertain reward or loss in bipolar versus major depression. Bipolar Disord. 2013 Dec;15(8):839-854. doi: 10.1111/bdi.12132. Epub 2013 Oct 21. PMID 24148027
- See also: An fMRI study of emotional face processing in adolescent major depression — https://doi.org/10.1016/j.jad.2014.06.037
- See also: A comparison between voxel-based cortical thickness and voxel-based morphometry in normal aging — https://doi.org/10.1016/j.neuroimage.2009.06.043